CLINICAL TRIAL: NCT05536882
Title: Randomized Controlled Trial Comparing the Efficacy of Adapalene 0.1% Gel to 10% Benzoyl Peroxide in Treating Molluscum Contagiosum.
Brief Title: MC RCT - BPO vs Adapalene
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The original PI left the institution prior to final IRB approval and the remaining study team did not have the resources to continue.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 14663
Record Dates: First submitted 2022-09-07; First posted 2022-09-13 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Molluscum Contagiosum
Keywords: /drug ther
MeSH Terms: conditions — Molluscum Contagiosum | interventions — Benzoyl Peroxide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benzoyl peroxide (Experimental): topical benzoyl peroxide 10% (vehicle choice per patient preference) applied 1-2x daily as tolerated until complete clearance or 12 week follow up
  Interventions: Drug: Benzoyl peroxide
- Adapalene (Active Comparator): adapalene 0.1% gel applied 1-2x daily as tolerated until complete clearance or 12 week follow up
  Interventions: Drug: Adapalene Gel

INTERVENTIONS:
Drug: Benzoyl peroxide — See arm description
  Arms: Benzoyl peroxide
Drug: Adapalene Gel — See arm description
  Arms: Adapalene

SUMMARY:
Non-blinded randomized controlled trial comparing efficacy of topical benzoyl peroxide 10% (vehicle choice per patient preference: e.g. gel, cream, lotion, wash) to topical adapalene 0.1% gel in the treatment of molluscum contagiosum in children aged 1 year old to 14 years old.

* Two treatment wings: topical benzoyl peroxide 10% (vehicle choice per patient preference) applied 1-2x daily as tolerated vs adapalene 0.1% gel applied 1-2x daily as tolerated.
* Primary outcome: Complete clearance at 12wks (defined as lack of identifiable papular molluscum contagiosum lesions on physical exam)
* Secondary outcomes: % change in lesion count at 12wks.

DETAILED DESCRIPTION:
* During the course of their normal workday, OU dermatology faculty and residents will be responsible for identifying and recruiting treatment-naïve patients being seen at the OU dermatology clinic for the diagnosis of molluscum contagiosum. These same faculty and residents will be responsible for approaching these patients regarding participation in the study. Chart review will not be a part of this selection process aside from what would naturally be done in the course of the patients' care. The same faculty and residents would be responsible for explaining the risks and benefits of study participation, obtaining written consent for study participation from a parent or guardian, obtaining verbal assent from patients aged 7-14 years old (as well as written assent for those capable of reading/writing), and randomizing patients to respective treatment wings using an online random number generator.
* # of MC lesions counted at time of recruitment, re-assessed at single follow up appointment at 12wks
* List of enrolled patients kept in excel spreadsheet on encrypted department shared drive. Data points added alongside patient names until all data points collected for an individual patient, then identifying information removed and replaced with a study number which will be used to refer to their de-identified data set going forward.
* Patients/caregivers would be responsible for obtainment and application of respective medications (both medications available over the counter for < $15)
* Primary and secondary outcomes will be assessed via Chi-square test

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 year to 14 years old seen in an OU Dermatology resident or faculty clinic and diagnosed with molluscum contagiosum who have not received prior treatment for this condition, and whose parent/guardian(s) desire treatment for this condition.

Exclusion Criteria:

* Patients who have received prior treatment for molluscum contagiosum.
* Patients with a history of adverse reaction to any topical retinoid, benzoyl peroxide, cinnamon, or other benzoic derivatives (e.g., salicylic acid, hydroquinone, catechol, vanillin).
* Pregnant females.
* Patients with caregivers who do not speak English.
* Patients with caregivers who are unable to provide consent.
* Patients who decline to assent for participation.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-09 (Actual)

PRIMARY OUTCOMES:
Complete clearance at 12 weeks | 12 weeks
  Defined as lack of identifiable papular molluscum contagiosum lesions on physical exam at 12 week follow up visit

SECONDARY OUTCOMES:
% change in lesion count at 12 weeks | 12 weeks

OTHER OUTCOMES:
Incidence and severity of irritant contact dermatitis and other adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hirshburg, MD, Principal Investigator — University of Oklahoma
Locations (1):
- OU Health Department of Dermatology, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saryazdi, S. The Comparative Efficancy of Benzoyl Peroxide 10% Cream and Tretinoin 0.05% Cream In The Treatment of Molluscum Contagiosum. Pediatric Derm. 2004, Vol. 20, 3, p. 399.
- [Background] Gupta, M. Adapalene in management of molluscum contagiosum in pediatric population. Our Dermatology Online. 2019, Vol. 10, 4, pp. 391-392.
- [Background] Kashif M, Tahir R, Hussain I. Efficacy and safety of trichloroacetic acid 35% versus adapalene 0.1% in treatment of molluscum contagiosum in children. Journal of Pakistan Association of Dermatologists. 2016, Vol. 26, 4, pp. 366-370.
- [Background] Na G, et al. P074 Clinical experience of adapalene on molluscum contagiosum. 프로그램북(구 초록집). 2016;68(2):373-373.
- [Background] Scheinfeld N. Treatment of molluscum contagiosum: a brief review and discussion of a case successfully treated with adapelene. Dermatol Online J. 2007 Jul 13;13(3):15. PMID 18328209
- [Background] Rajouria EA, Amatya A, Karn D. Comparative study of 5 % potassium hydroxide solution versus 0.05% tretinoin cream for Molluscum Contagiosum in children. Kathmandu Univ Med J (KUMJ). 2011 Oct-Dec;9(36):291-4. doi: 10.3126/kumj.v9i4.6347. PMID 22710541
- [Background] Kim MS, Chun DK, Lee YS, et al. Treatment of Molluscum Contagiosum with Topical Tretinoin Therapy. Korean J Dermatol. 2001;39(6):666-670.